CLINICAL TRIAL: NCT07068230
Title: Comparing the Effects of Ondansetron Versus Dexamethasone on the Incidence of Post-dural Puncture Headache (PDPH) , Nausea and Vomiting After Spinal Anaesthesia of Parturients Undergoing Caesarean Section.
Brief Title: Ondansetron and Dexamethasone for Prevention of PDPH, Nausea, and Vomiting
Acronym: PDPH-N/V
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Minia University (Other)
Collaborators: Faculty of Medicine, Minia University (Unknown)
Responsible Party: Principal Investigator, Mokhtar Mostafa Mahran Mohamed, lecture, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EMUH-PDPH-2018-001; research ethical committee (Other: faculty of medicine, minia university)
Record Dates: First submitted 2025-07-06; First posted 2025-07-16 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Postdural Puncture Headache; Postoperative Nausea and Vomiting; Obstetric Anesthesia Problems
Keywords: Ondansetron; Dexamethasone; Postdural Puncture Headache; Nausea; Vomiting
MeSH Terms: conditions — Post-Dural Puncture Headache; Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — Ondansetron; Dexamethasone; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: This study is a parallel assignment model in which 150 parturients undergoing elective cesarean section under spinal anesthesia were randomized into three groups in a 1:1:1 ratio to receive either intravenous ondansetron, dexamethasone, or placebo. Each participant was assigned to one intervention group and remained in that group for the duration of the study.
Who Masked: Participant, Care Provider
Masking Description: This was a double-blind study. Both the patients and the care providers (anesthesiologists) were blinded to the group assignments. Study medications were prepared in identical 5 mL syringes labeled A, B, or C by an independent supervisor who was not involved in patient care, drug administration, or data collection. Neither the participants nor the medical staff administering the anesthesia or assessing outcomes were aware of the group allocations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ondansetron Group (Experimental): Participants in this group received 8 mg of intravenous ondansetron diluted to 5 mL with normal saline, administered 5 minutes before spinal anesthesia.
  Interventions: Drug: Ondansetron 8mg
- Dexamethasone Group (Experimental): Participants in this group received 8 mg of intravenous dexamethasone diluted to 5 mL with normal saline, administered 5 minutes before spinal anesthesia.
  Interventions: Drug: Dexamethasone
- Placebo Group (Experimental): Participants in this group received 5 mL of intravenous normal saline as placebo, administered 5 minutes before spinal anesthesia.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ondansetron 8mg — Ondansetron 8 mg IV Administered 5 minutes before spinal anesthesia
  Other Names: zofran
  Arms: Ondansetron Group
Drug: Dexamethasone — Dexamethasone 8 mg IV Administered 5 minutes before spinal anesthesia
  Arms: Dexamethasone Group
Drug: Saline — 5ml normal saline Administered 5 minutes before spinal anesthesia
  Other Names: normal saline
  Arms: Placebo Group

SUMMARY:
This prospective, randomized, double-blind, placebo-controlled study was conducted at the Obstetrics and Gynecology Department of El-Minia University Hospital from October 2018 to October 2019. It enrolled 150 parturients aged 18-45 years undergoing elective cesarean section under spinal anesthesia. Participants were randomly assigned to one of three groups to receive either 8 mg IV ondansetron, 8 mg IV dexamethasone, or 5 mL of IV normal saline 5 minutes before spinal anesthesia. The primary objective was to evaluate the effectiveness of prophylactic ondansetron and dexamethasone in reducing the incidence of postdural puncture headache (PDPH). Secondary outcomes included severity and duration of PDPH, incidence and severity of nausea and vomiting, hemodynamic parameters, and neonatal Apgar scores. Ethical approval was obtained and verbal informed consent was collected from all participants.

DETAILED DESCRIPTION:
This study is a single-center, prospective, randomized, double-blind, placebo-controlled clinical trial conducted to evaluate the efficacy of prophylactic intravenous administration of ondansetron and dexamethasone in reducing the incidence and severity of postdural puncture headache (PDPH), and postoperative nausea and vomiting (PONV), in parturients undergoing elective cesarean section under spinal anesthesia.

A total of 150 parturients (ASA I or II), scheduled for cesarean delivery at Minia University Hospital, were randomly allocated into three parallel groups (1:1:1 ratio) using computer-generated randomization with sealed opaque envelopes to conceal allocation.

All patients received standard spinal anesthesia with 0.5% hyperbaric bupivacaine via a 25-gauge Quincke spinal needle in the sitting position at the L3-L4 or L4-L5 interspace. Prior to spinal anesthesia, patients in:

Group A (Ondansetron group) received 8 mg ondansetron IV (diluted to 5 mL in saline),

Group B (Dexamethasone group) received 8 mg dexamethasone IV (diluted to 5 mL),

Group C (Control group) received 5 mL of 0.9% normal saline IV.

Study drugs were administered 5 minutes prior to the intrathecal injection. Blinding was maintained for patients, anesthesiologists, and outcome assessors.

PDPH was assessed for 7 days postoperatively. A standardized questionnaire and the Corbey scale were used to evaluate headache onset, severity, duration, and need for analgesics. Nausea and vomiting were assessed intraoperatively and postoperatively (up to 48 hours). Standard antiemetic rescue therapy was available as needed.

The protocol adhered to CONSORT guidelines and was approved by the Minia University Faculty of Medicine Research Ethics Committee. All participants provided written informed consent prior to enrollment.

This trial investigates whether prophylactic ondansetron or dexamethasone, individually, can significantly reduce PDPH and PONV compared to placebo. The results are expected to inform perioperative management and enhance maternal outcomes in cesarean section under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria

* Female patients aged 18 to 45 years
* Body Mass Index (BMI) between 23-27 kg/m²
* American Society of Anesthesiologists (ASA) physical status I or II
* Scheduled for elective cesarean section under spinal anesthesia Exclusion Criteria
* Refusal to participate
* Conversion to general anesthesia due to failed spinal block
* Known hypersensitivity to ondansetron or dexamethasone
* Contraindications to study medications, including:

  * Diabetes mellitus
  * Active infection
  * Prolonged QT interval
* History of tobacco or drug use
* Coagulopathy or localized infection at the spinal injection site
* High-risk pregnancy (e.g., preeclampsia, placenta previa)
* History of chronic headache or migraine

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females of childbearing age undergoing elective cesarean section under spinal anesthesia
Enrollment: 150 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Postdural Puncture Headache (PDPH) | Up to 14 days postoperatively
  The primary outcome is the proportion of participants in each group who develop postdural puncture headache within 14 days following spinal anesthesia for elective cesarean section. Diagnosis is based on clinical criteria assessed during follow-up calls on postoperative days 7 and 14 by a blinded anesthesiologist.

SECONDARY OUTCOMES:
Severity of PDPH | Up to 14 days postoperatively
  Severity of PDPH will be assessed using the Corbey Headache Severity Scale, which categorizes headache as:
  Mild (no limitation of daily activity),
  Moderate (some limitation of activity but no bed rest required), and
  Severe (requires bed rest). Scale: Mild to Severe - higher levels indicate worse outcome
Duration of PDPH | Up to 14 days postoperatively
  Duration (in days) from onset to resolution of PDPH symptoms in affected participants.
Incidence of Nausea and Vomiting (N/V) | Intraoperatively and up to 4 days postoperatively
  Incidence of intraoperative and postoperative nausea and vomiting, assessed using a 4-point scale (0 = none, 1 = nausea only, 2 = nausea and vomiting, 3 = repeated vomiting).
Neonatal Outcome (Apgar Score at 1 and 5 minutes) | At 1 minute and 5 minutes after birth
  Neonatal wellbeing will be assessed using the Apgar Score, a standardized clinical scale that evaluates Appearance (skin color), Pulse (heart rate), Grimace (reflex irritability), Activity (muscle tone), and Respiration.
  Scale Description:
  Minimum Score: 0 (worst outcome)
  Maximum Score: 10 (best outcome)
  Higher scores reflect better neonatal condition

CONTACTS AND LOCATIONS:
Overall Officials: mokhtar m mohamed, MD, Principal Investigator — El-Minia University Hospital
Locations (1):
- El-Minia University Hospital, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to primary and secondary outcomes will be made available upon reasonable request from qualified researchers for academic purposes. Data will be shared beginning 6 months after publication and available for up to 2 years.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be available beginning 6 months after publication and ending 2 years after publication
Access Criteria: Data will be available to qualified researchers whose proposed use of the data has been approved by an independent review committee. Requests should be directed to the principal investigator via institutional contact.